CLINICAL TRIAL: NCT07368231
Title: Forest Therapy and Mindfulness in Highly Sensitive Persons (HSP): A Multicenter Randomized Interventional Study Over Approximately 22 Weeks
Brief Title: Forest Therapy and Mindfulness for Highly Sensitive Persons
Acronym: HSP-FOREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IFM International Forest Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSP-FOREST-2025-RTC-C; HSP-FOREST-2025-C (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2025-12-12; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Stress (Psychology); Well-Being, Psychological; Mind-Body Therapies; Complementary Therapies; Mindfulness; Preventive Medicine
Keywords: Forest Bathing; Forest Therapy; Shinrin Yoku; Mindfulness; Forest Medicine; Highly Sensitive Person (HSP); Stress reduction; Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Forest Therapy; Mindfulness; Psychotherapy; Reproductive Techniques, Assisted; Aromatherapy

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group interventional study in which participants are assigned in a 1:1 ratio to one of two arms: a forest therapy plus mindfulness intervention or an active indoor sensory control condition. Participants remain in their assigned arm for the full duration of the study.
Who Masked: Outcomes Assessor
Masking Description: Due to the behavioral nature of the interventions, participants and care providers are not blinded. Outcome assessors are masked to group allocation during data collection and evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forest Therapy + Mindfulness + Psychotherapy (Experimental): Participants will undergo an approximately 22-week program with 4.5 hours weekly in forest settings. Sessions include a guided forest walk, mindfulness meditation, structured sensory awareness exercises, facilitated group reflection, and a brief psychotherapeutic component focused on emotional processing and cognitive regulation. Intervention delivery is standardized through facilitator training and a predefined session manual.
  Interventions: Behavioral: Forest Therapy + Mindfulness + Psychotherapy
- Indoor Sensory Control (Art and Aromatherapy) (Active Comparator): Structured indoor sensory-based group sessions delivered weekly over approximately 22 weeks. Sessions are designed to match the experimental intervention in duration, structure, facilitator contact, and social interaction, without exposure to forest or outdoor natural environments. Activities include creative tasks, guided aromatherapy, sensory-focused exercises, and facilitated group discussion according to a predefined protocol.
  Interventions: Behavioral: Behavioral: Indoor Sensory Control (Art and Aromatherapy)

INTERVENTIONS:
Behavioral: Forest Therapy + Mindfulness + Psychotherapy — Participants will undergo a approximately 22-week program with 4.5 hours weekly in forest settings. Each session includes:
  A 2-hour guided walk with scheduled rest/hydration breaks
  Mindfulness meditation (20-30 minutes)
  Discussion/reflection segment (~20 minutes) for participants to express sensations, experiences, or doubts
  A psychotherapeutic component focused on emotional processing and cognitive regulation
  Sensory observation (5-10 minutes) of forest stimuli (olfactory, auditory, tactile, visual)
  Post-session journaling capturing emotional and sensory feedback
  Monitoring of environmental parameters (temperature, humidity, wind, estimated phytoncide levels)
  Standardized facilitator training and session protocols to ensure consistency across sites
  This protocol is distinguished by integrating forest immersion, mindfulness, psychotherapy, and sensory training in a unified intervention tailored for Highly Sensitive Persons (HSP).
  Arms: Forest Therapy + Mindfulness + Psychotherapy
Behavioral: Behavioral: Indoor Sensory Control (Art and Aromatherapy) — Structured indoor sensory-based group sessions delivered weekly over approximately 22 weeks. Activities include creative tasks, guided aromatherapy, and sensory-focused exercises conducted in indoor, non-forest environments. Sessions are designed to match the experimental intervention in duration, structure, facilitator contact, and social interaction, according to a predefined protocol.
  Arms: Indoor Sensory Control (Art and Aromatherapy)

SUMMARY:
This randomized, multicenter interventional study evaluates a combined forest therapy (shinrin-yoku) and mindfulness-based program in adults with high sensory-processing sensitivity confirmed using a validated instrument. Participants are randomized (1:1) to either a forest-based intervention or an active indoor sensory control condition. The intervention is delivered over approximately 22 weeks according to a predefined protocol, with assessments conducted at baseline and at the end of the intervention.

DETAILED DESCRIPTION:
This is a multicenter, randomized, parallel-group interventional study in adults with high sensory-processing sensitivity confirmed using a validated instrument. Participants are randomized 1:1 to one of two study arms at study entry and remain in their assigned group for the duration of the study.

Intervention delivery is standardized across participating sites through facilitator training and a predefined session manual. The experimental arm consists of structured sessions conducted in forest environments and includes guided walking, mindfulness-based practices, and structured sensory awareness activities, with facilitated group reflection. The active comparator arm consists of structured indoor group activities designed to match the experimental arm in duration, group interaction, and facilitator contact, without exposure to forest or outdoor natural environments.

Study procedures and assessment schedules are predefined in the protocol and implemented in accordance with applicable ethical requirements and Good Clinical Practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* High sensory-processing sensitivity confirmed using a validated instrument (e.g., HSPS/Aron scale)
* Able to perform moderate physical activity (e.g., walking)
* Able to provide written informed consent

Exclusion Criteria:

* Severe psychiatric disorder or acute clinical instability
* Medical condition contraindicating moderate physical activity
* Use of medications with strong autonomic or neuroendocrine effects (e.g., high-dose systemic corticosteroids; selected beta-blockers)
* Recent participation in a structured mindfulness or forest-therapy program
* Pregnancy or unstable medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Score (PSS-10) From Baseline to End of Intervention | Baseline to end of intervention (approximately 22 weeks)
  Measure the difference in total score on the Perceived Stress Scale (PSS-10) between baseline and the end of the intervention. PSS-10 comprises 10 items scored 0-40, with higher scores indicating greater perceived stress.

SECONDARY OUTCOMES:
Change in Psychological Well-Being Score (WHO-5) From Baseline to End of Intervention | Baseline to end of intervention (approximately 22 weeks)
  Measure the difference in total score on the WHO-5 Well-Being Index between baseline and the end of the intervention. WHO-5 comprises 5 items scored 0-25, with higher scores indicating better well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Ana I Sánchez Hdz, Principal Investigator — IFM International Forest Medicine
Locations (2):
- Spain (2):
  - IFM International Forest Medicine, Ronda, Andalusia
  - Sessions conducted in natural forest settings within the Serranía de Ronda, specifically the Valle del Genal area, Ronda, Andalusia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data supporting publications arising from this study will be shared with qualified researchers beginning 6 to 36 months after publication.
Supporting Information: Study Protocol
Time Frame: Beginning 6 months after publication and available for up to 36 months.
Access Criteria: Access will be granted to qualified researchers upon reasonable request, subject to approval by the responsible ethics committee and execution of a data use agreement. Requests must include a research proposal and analysis plan.

REFERENCES:
- [Result] Sánchez Hdz, Ana I. Forest Therapy and Mindfulness in Highly Sensitive Persons (HSP): Confirmatory Evidence from a Multicenter Randomized Controlled Trial with 6-Month Follow-up. Zenodo. DOI: 10.5281/zenodo.17361382. Available at: https://zenodo.org/records/17361382
- See also: Forest Therapy and Mindfulness for Stress Reduction and Well-being in Highly Sensitive Persons (Pilot RCT)" (HSP-FOREST) — https://clinicaltrials.gov/study/NCT07183917
- Available data/document: Study Protocol: ZENODO17361382 — https://zenodo.org/records/17361382 — Access via the URL provided (Zenodo record)